CLINICAL TRIAL: NCT01813799
Title: A Multicenter, Placebo-controlled, Randomized, Double-blind, Phase II Clinical Trial With Diabetic Neuropathy Patients is Designed to Evaluate the Safety and Efficacy of the DA-9801 Tablet for Neuropathic Pain and to Decide Optimal Dose.
Brief Title: Study of DA-9801 to Treat Diabetic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA9801_DN_II
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — DA-9801

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DA-9801 300mg (Experimental)
  Interventions: Drug: DA-9801 300mg
- DA-9801 600mg (Experimental)
  Interventions: Drug: DA-9801 600mg
- DA-9801 900mg (Experimental)
  Interventions: Drug: DA-9801 900mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-9801 300mg — 300mg of DA-9801 tablet is assigned at week 0 point and is taken for 8 continuous weeks, 3 times a day.
  Arms: DA-9801 300mg
Drug: DA-9801 600mg — 600mg of DA-9801 tablet is assigned at week 0 point and is taken for 8 continuous weeks, 3 times a day.
  Arms: DA-9801 600mg
Drug: DA-9801 900mg — 900mg of DA-9801 tablet is assigned at week 0 point and is taken for 8 continuous weeks, 3 times a day.
  Arms: DA-9801 900mg
Drug: Placebo — Placebo is assigned at week 0 point and is taken for 8 continuous weeks, 3 times a day.
  Arms: Placebo

SUMMARY:
This is a Phase II dose-ranging study to evaluate the effectiveness and safety of DA-9801 in the treatment of pain associated with diabetic neuropathy. Subjects will receive either 300mg, 600mg, 900mg or placebo, three times daily for eight weeks. During treatment, pain score by Likert numerical rating scale, Patient Global Impression of Improvement (PGI-I) and Change in Clinical Global Impression(CGI)are accessed to evaluate the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* the age of 20 ~ 70
* Type I or Type II Diabetes
* HbA1c ≤11%
* Patients with diabetic neuropathic pain for at least 3 months
* Patients corresponding to average pain level of 4 points or more for 24 hours evaluated with 11-point Likert scale

Exclusion Criteria:

* neuropathic pain due to other causes or another stronger pain other than neuropathic pain
* abnormal in blood pressure, weight, ALT/AST, Serum creatinine
* positive reaction in HIV, HBV, or HCV
* experience of suicide try or Mental Illness Medical History
* BDI(Beck Depression Inventory) grade exceeding 21 points chronic alcohol abuse history

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Difference in average 24-h pain intensity (Likert scale) between before and after IP administration | 8 weeks
  Subject records the average pain intensity for the past 24 hours in the patient diary at the same time every morning.

SECONDARY OUTCOMES:
Inter-group difference in average 24-h pain intensity (Likert scale) | 8 weeks
  The mean value of the last one week since the date of visit was calculated to compare the difference between treatment groups.
Most severe mean pain intensity (Likert Scale) | 4, 8 weeks
  Subject records the most severe pain intensity for the past 24 hours in the patient diary at the same time every morning.
Overnight pain intensity (Likert Scale) | 4, 8 weeks
  Subject records the overnight pain intensity during the previous night in the patient diary at the same time every morning.
Patient's Global Impression of improvement (1 point ~ 7 point) | 4, 8 weeks
  Subject evaluated the level of symptom improvement during the visits after IP administration.
Clinical Global Impression of severity (1 point ~ 7 point) | 4, 8 weeks
  Investigator evaluated the level of symptom severity when a subject visited the institution.
Average daily dose of acetaminophen | everyday(-2 weeks~0), everyday(0~8 weeks)
  Subject records dose of acetaminophen during the past 24 hours in patient diary at the same time every

CONTACTS AND LOCATIONS:
Overall Officials: Bongyeon Cha, M.D., Principal Investigator — The Catholic University of Korea; Hyeok Sang Gwon, M.D., Principal Investigator — Catholic University Yeouido St. Mary's Hopspital; Inkyung Jeong, M.D., Principal Investigator — Gangdong Kyunghee University Hospital; Ji Hyeon Lee, M.D., Principal Investigator — Daegu Catholic University Medical Center; Jeong Guk Kim, M.D., Principal Investigator — Kyungpook National University Hospital; In Ju Kim, M.D., Principal Investigator — Busan National University Hospital; Young Min Cho, M.D., Principal Investigator — Seoul National University Hospital; Chun Hee Jung, M.D., Principal Investigator — Yonsei University Wonju Christian Hospital; Jyeong Hyeon Park, M.D., Principal Investigator — Inje University; Mun Seok Nam, M.D., Principal Investigator — Inha University Hospital; Dong Hyeok Cho, M.D., Principal Investigator — Chonnam National University Hospital; Min Kyong Moon, M.D., Principal Investigator — SMG-SNU Boramae Medical Center; Chong Hwa Kim, M.D., Principal Investigator — Sejong General Hospital; Kwan Pyo Ko, M.D., Principal Investigator — Jeju National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea